CLINICAL TRIAL: NCT00565175
Title: Histamine H2 Antagonism as Adjuvant Therapy in Treatment Resistant Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jesper Ekelund (Other)
Collaborators: Finland: Lilly saatio foundation (Unknown)
Responsible Party: Sponsor-Investigator, Jesper Ekelund, Professor of psychiatry, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-006636-22; 2006-006636-22 (EudraCT Number)
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
Keywords: Treatment resistant; Chronic
MeSH Terms: conditions — Schizophrenia; Bronchiolitis Obliterans Syndrome | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- famotidine (Experimental)
  Interventions: Drug: famotidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Microcrystallized cellulose)

INTERVENTIONS:
Drug: famotidine — Capsules containing 100 mg of famotidine p.o., twice daily for 4 weeks.
  Other Names: Famotidin Hexal
  Arms: famotidine
Drug: Placebo (Microcrystallized cellulose) — Placebo administered in identical capsules as the experimental drug.
  Other Names: Microcrystallized cellulose
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate whether blockade of the histamine H2 receptors in the brain will have any beneficial effect on the symptoms of subjects with schizophrenia.

DETAILED DESCRIPTION:
Histamine functions as a neurotransmitter in the brain. It has an important role as modulator of the release of other neurotransmitters, including dopamine.

The histamine receptors are widely expressed in the brain, H1 and H2 receptors are post-synaptic, H3 a pre-synaptic autoreceptor. There is an abundance of neurobiologic data from animal and human studies supporting the role of histamine in the pathogenesis and treatment of psychoses.

In 1990 a case report of a treatment resistant subject with schizophrenia whos symptoms improved markedly when he was prescribed a H2 antagonist because of peptic ulcer. Later, a open-label trial including 18 patients has been performed, reporting significant symptom reduction, especially on negative symptoms. Also the subjective comments both by the subjects and the investigators in that study were optimistic and suggested an effect primarily on negative symptoms.

The present study will be the first double-blind, randomized, placebo controlled, parallel group study of the subject matter. The study focuses on treatment resistant schizophrenia cases in the stable phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia assessed by SCID-I (DSM-IV) as well as RDC-criteria
* Patient record mention of schizophrenia (ICD-10) at least 5 years previously
* Disability pension due to psychiatric disorder
* At least 3 points on the CGI scale

Exclusion Criteria:

* Epilepsy or a history of unclear seizures
* Stroke
* Parkinson's disease
* AIDS
* Substance addiction or abuse within 3 months prior to enrolment.
* Individuals who are deemed at risk for aggressive behavior or suicide by their clinician
* Pregnant and breast-feeding subjects
* Serious unstable physical illness
* Persons who have been deemed legally incapacitated according to Finnish law (Laki holhoustoimesta 1.4.1999/442, 3. luku, 18 §)
* Individuals who use H2-antagonists as prescribed by a physician
* Known allergy to famotidine or any other component of the Pepcidin® 40 mg tablet
* Glomerular Filtration Rate (GFR) according to the Cockcroft-Gault formula < 30 ml/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Negative Symptoms (SANS) score | 5 weeks

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) score | 5 weeks
Clinical Global Impression (CGI) score | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Ekelund, MD-PhD, Principal Investigator — Helsinki University Central Hospital
Locations (5):
- Finland (5):
  - HUCH Department of Psychiatry, Helsinki
  - Kellokosken sairaala, Kellokoski
  - Lohjan sairaanhoitoalue, Lohja
  - Vaasa Hospital District, Vaasa
  - Peijaksen sairaala, Vantaa

REFERENCES:
- [Derived] Meskanen K, Ekelund H, Laitinen J, Neuvonen PJ, Haukka J, Panula P, Ekelund J. A randomized clinical trial of histamine 2 receptor antagonism in treatment-resistant schizophrenia. J Clin Psychopharmacol. 2013 Aug;33(4):472-8. doi: 10.1097/JCP.0b013e3182970490. PMID 23764683